CLINICAL TRIAL: NCT06277232
Title: Developing an Innovative EHealth Intervention to Support Patients' Nutrition Care During Pain Rehabilitation - a Feasibility and Pilot Study
Brief Title: Nutrition Care in Patients Living with Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ostergotland County Council, Sweden (Other); Swedish Fibromyalgia syndrome association (Unknown)
Responsible Party: Principal Investigator, Huan-Ji Dong, MD, PhD, Associate Professor (Docent), Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMV-2023-00504; 2022-05364-02 (Other: The Swedish Ethical Review Authority)
Record Dates: First submitted 2024-02-03; First posted 2024-02-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-08

CONDITIONS: Nutrition Poor; Overweight and Obesity; Mobile Phone Use; Pain, Chronic
Keywords: Chronic pain; Nutrition care; Pain rehabilitation; eHealth
MeSH Terms: conditions — Malnutrition; Overweight; Obesity; Cell Phone Use; Chronic Pain | interventions — Nutrition Therapy; Educational Status; Cognitive Behavioral Therapy; Relaxation Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Repeated measures, single-subject withdrawal design. All subjects who enroll in the study will receive the intervention and there is no randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Other): Through the Diet4painrelief platform, the dietician will follow up the progress of each participant in different timepoints during pain rehabilitation process: 4 weeks before the Interdisciplinary Pain Rehabilitation Program (IPRP), 1-2 meetings with patients as well as other professionals integrated in IPRP, and 4 weeks after IPRP rehabilitation (via chat function).
  The IPRP is conducted in groups of six to nine participants and is based on cognitive behavioral treatment principles and included physiotherapy, ergonomics, training in coping strategies, occupational therapy, and education in pain management. An IPRP delivers a group-treatment format by an interdisciplinary team (i.e., physician in rehabilitation, a physiotherapist, an occupational therapist, and a psychologist). The IPRP lasts for 12 weeks.
  Interventions: Other: Nutrition care; Behavioral: Dialogue and education (part of Interdisciplinary Pain Rehabilitation Program); Behavioral: activity training (part of Interdisciplinary Pain Rehabilitation Program); Behavioral: meetings (part of Interdisciplinary Pain Rehabilitation Program); Behavioral: Cognitive behavioral therapy (part of Interdisciplinary Pain Rehabilitation Program); Behavioral: Relaxation techniques (part of Interdisciplinary Pain Rehabilitation Program); Behavioral: Physical exercise (part of Interdisciplinary Pain Rehabilitation Program)

INTERVENTIONS:
Other: Nutrition care — Nutrition care is designed to include nutrition assessment (e.g., malnutrition screening, monitoring weight changes, etc.), optimization of individual dietary patterns, and evaluation. Through the Diet4painrelief platform, a dietician will follow up the progress of each participant in different timepoints and also plan meetings with other professionals in IPRP. A dietitian together with a physician in rehabilitation are responsible for the administration of the procedure.
Behavioral: Dialogue and education (part of Interdisciplinary Pain Rehabilitation Program) — Dialogue and education consists of patient education, training in wellness and healthy living habits, meetings with families, video feedback, and couples therapy and self-training (e.g., home lessons, activity diary, physical self-training, reflection time, and self-analysis. . In addition, lectures in basic pain science and pain management are offered for both patients as well as for relatives, friends, and colleagues.
Behavioral: activity training (part of Interdisciplinary Pain Rehabilitation Program) — Activity training includes graded activity training, and exposure training, which are delivered by an interdisciplinary team (i.e., a physiotherapist, an occupational therapist, and a psychologist).
Behavioral: meetings (part of Interdisciplinary Pain Rehabilitation Program) — The meetings consist of conferences with patients, rehabilitation team, vocational guidance, rehabilitation coordinator, goal-setting meetings, and meetings to check goal achievement.
Behavioral: Cognitive behavioral therapy (part of Interdisciplinary Pain Rehabilitation Program) — Acceptance and Commitment Therapy (ACT, e.g., goal compass, training in ACT principles, and mindfulness) is mainly delivered by psychologist in a group-treatment (e.g., training in coping strategies). The cognitive behavioral principles are also used in physiotherapy, ergonomics, and education in pain management.
Behavioral: Relaxation techniques (part of Interdisciplinary Pain Rehabilitation Program) — This group-treatment is mainly format by a physiotherapist and psychologist in an interdisciplinary team.
Behavioral: Physical exercise (part of Interdisciplinary Pain Rehabilitation Program) — This group-treatment is mainly format by a physiotherapist in an interdisciplinary team.

SUMMARY:
The investigators' purpose is to develop and test the feasibility, usability, and satisfaction of the Diet4painrelief app as a platform for implementing nutrition care in a specialist pain rehabilitation clinic. The Diet4painrelief will consist of two components: a) a screening tool for nutrition status b) an individually tailored behavior change program aiming to improve the dietary habits and behaviors of patients living with chronic pain.

The study is planned to include 20 patients with complex chronic pain and non-optimal BMI (underweight or overweight/obesity) to examine the feasibility and outcomes of evidence-based Interdisciplinary Pain Rehabilitation Program (IPRP) integrated with nutrition care. The Diet4painrelief includes a screening tool to assess basic nutritional status as well as their intake of key unhealthy and healthy foods and drinks (through three 24hour-dietary recordings or food diary). Thereafter, the patients receive a personalized behavior change program for dietary optimization. The investigators will design and adapt 6 modules in the digital platform (Diet4painrelief app) based on the International Association for the Study of Pain (IASP) recommendations (6 aspects about 'nutrition and pain') and Sweden's food culture. Clinical outcomes using patient-reported data on socio-demographics, pain aspects, psychometric data, physical disability, and quality of life will be measured at three occasions: first appointment (Pre-IPRP), immediately after completing the rehabilitation program (Post-IPRP), and at a 12-month follow-up (FU-IPRP). Blood samples will be taken to identify biomarkers at the same occasions that provide objective information on metabolic and nutritional abnormalities and further to evaluate the effect of the dietary intervention on changing of pain rehabilitation outcomes.

DETAILED DESCRIPTION:
Potential participants are patients referred to a specialized pain and rehabilitation clinic due to complex chronic non-malignant pain conditions. A bio-psycho-social assessment revealed that these patients presented psychological symptoms and other comorbidities, reported large difficulties with their pain, and their condition severely affected their working life and participation in social activities. They often did not respond to routine pharmacological/ physiotherapeutic treatments delivered in a mono-disciplinary fashion. The potential participants received written information about the Swedish Quality Registry for Pain Rehabilitation (SQRP) (www.ucr.uu.se/nrs/) research and gave their written consent. The SQRP is mainly based on patient reported outcome measures (PROM) about socio-demographics, pain aspects, body weight and height, psychometric data, physical disability, and quality of life. Patients will complete the questionnaires of SQRP on three occasions: (1) before assessment on the first visit to the clinic (baseline or Pre-IPRP); (2) immediately after IPRPs (Post-IPRP); and (3) at the 12-month follow-up after IPRP discharge (FU-IPRP). Information on body height and weight were self-reported or measured and registered during the clinical assessment. All patients who respond to SQRP and have a Body Mass Index (BMI) ≥ 25 kg/m2 will be asked to participate in the study and may submit blood samples (see below).

After completing the informed consent to participate, the participants will fill out a food diary. For those who fail to complete food diaries, a dietician will book an individual meeting to go through three 24hour-dietary recordings. They will be introduced to get access to Diet4painrelief app by one research assistant. One dietician will make individualized plans of nutrition care in the app based on the information from the screening (through three 24hour-dietary recordings or food diary). The patient will receive dietary recommendations based on each patient's need for nutrition. The investigators will design and adapt 6 modules in the digital platform (Diet4painrelief app) based on the IASP recommendations (6 aspects about 'nutrition and pain') and Sweden's food culture. Overall, the app consists of the several features: weekly, push notifications, self-monitoring and feedback features of pain, diet, and recipe feature. The users will receive a text message prompting a brief weekly screening of the nutrition aspects, followed by feedback on individual screening results in comparison with recommendations they initially have received from the dietician. The feedback will be delivered on a graduated colored scale addressing diet aspects (agreement with recommendations). All users will then access a personal interactive dashboard with pictures representing nutritional behavior.

Through the Diet4painrelief platform, the dietician will follow up the progress of each participant in different timepoints during pain rehabilitation process: 4 weeks before standard pain rehabilitation program, 1-2 meetings integrated in rehabilitation process, and 4 weeks after the rehabilitation (via chat function). Participants' perceptions of using eHealth (digital healthcare applications) will be evaluated through individual interviews with the valid questionnaires (personal feelings, utility, and technical issues).

Blood samples will be collected in P100 tubes for all participants at Pre-IPRP, Post-IPRP and FU-IPRP. The sample will be centrifuged at 2500 g for 20 min at room temperature within 2-4 hours. Plasma will be extracted by carefully removing the upper part of the supernatant in fractions to a 10 mL tube, and after mixing gently will be aliquoted into 200 µl in 0.6 mL eppendorf tubes and stored at -86°C. The cell fraction will be removed to a new tube and stored at -86°C. The samples (marked with a code number) will be sent to the clinic´s research laboratory for centrifugation and storing in -86°C. The omic analysis aims to identify biomarkers that provide objective information on metabolic and nutritional abnormalities that can cause or worsen pain, further to objectively evaluate the effect of the dietary intervention on changing of pain rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self reported Body Mass Index (BMI)>=25;
* Written consent to participate and attend to the pain rehabilitation program due to disabling chronic pain (on sick leave or experiencing major interference in daily life due to chronic pain)
* Agreement not to participate in other parallel treatments for weight reduction
* Not currently using medications of weight reduction
* Available to get access to internet via own mobile/cellphone.

Exclusion Criteria:

* Health conditions such as pregnancy, active metabolic disease, rheumatoid arthritis, and serious psychiatric disease (investigator's judgement, eg, psychosis or suicidal ideation);
* Coagulation disorders with predisposition to bleeding, medication with anticoagulants (low- dose aspirin is permitted);
* hypersensitivity to anaesthetic
* Difficulties in understanding the Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (numeric rating scale) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up
  A numeric rating scale, 0=no pain, 10=worst pain experienced
Pain interference (one aspect in Multidimensional Pain inventory) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) ) and later at 12-month follow-up
  Multidimensional Pain inventory Swedish version is based on 11 items, each scored 0-6. To measure pain-related interference in everyday life, 0 = no interference, 6 = extreme interference
Dietary habits (a lifestyle questionnaire) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up
  A lifestyle questionnaire measures self-reported regular mealtime, frequency of vegetables and fruits intake, frequency of fast-food and confectionary consumption.
Perceived Usability (System Usability Scale) | Participants will be asked about their perceived benefit twice, after the rehabilitation (12 weeks) and later at 12-month follow-up.
  System Usability Scale (0-100) is composed of 10 statements that are scored on a 5-point scale of strength of agreement.
Perceived benefit (numeric rating scale) | Participants will be asked about their perceived benefit twice, after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Participants' opinions as to the benefits or effectiveness of the intervention are collected via an 11-point scale asking, "Overall, how beneficial was nutrition care for your pain? End points for the 11-point scale are: 0="Not beneficial at all" ; 10=Extremely beneficial". Participants are also asked to provide comment on whether they think additional treatment as provided in this study will improve nutrition care. A higher score suggests a greater self-perceived benefit.
Adherences/ compliances of nutritional care (numeric rating scale) | Participants will be asked about their perceived benefit twice, after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Regarding screening, diet recommendations and sustainable motivation for eating behavior changes. This patient adherence object score is a scale of 0-10 about "How well have you been following your diet plan? 0= not at all, 4= somewhat, and 10= following the plan very well. A higher score indicates a better adherence/compliance.

SECONDARY OUTCOMES:
Difficulty sleeping (Insomnia Severity Index) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Insomnia Severity Index (ISI, 0-28) consists of 7 items and each is scored 0-4. The score is divided into 4 categories: no clinically significant insomnia (ISI 0-7); sub-threshold insomnia (ISI 8-14); moderate clinical insomnia (ISI 15-21); and severe clinical insomnia (ISI 22-28).
Emotional distress (The Hospital Anxiety and Depression Scale, HAD) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Depression and Anxiety using Hospital Anxiety and Depression Scale (0-42). One subscale (depression or anxiety) has seven items with a scoring range of 0 to 21; the lower score indicates a lower possibility of anxiety or depression.
Impact of chronic pain (Multidimensional Pain inventory) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Multidimensional Pain inventory Swedish version- Life control (0-6) is based on 4 items, each scored 0-6. A higher score indicates a better control.
Health- related quality of life 1 (EQ-5D) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  EQ- 5D, Consists of two parts. The first part is an index obtained from five dimension items scored 0-5. The second part is self- estimation of today's health according to a 100- point thermometer- like scale (EQ5D- VAS) with defined end points (high values indicate better health and low values indicate worse health).
Health- related quality of life 2 (RAND-36) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  RAND- 36 (0-100), consists of 36 items in eight subcategories scored varying between 0 and 100% (with fixed intervals). The mean for each subscale is calculated
Pain coping (Chronic Pain Acceptance Questionnaire, CPAQ) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Chronic Pain Acceptance Questionnaire (CPAQ) is a 20item scale with 2 subscales: activity engagement independent of pain (score range 0-66; denoted CPAQ-engagement) and willingness to accept pain/need to control pain (score range 0-54; denoted CPAQ-willingness). All items are rated on a scale from 0 (never true) to 6 (always true). High values mirror high activity engagement and high pain willingness, respectively.
Fear of movement (Tampa scale for Kinesiophobia) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Tampa scale for Kinesiophobia (0-68),17 items, each scored 0-4 according to agreement with statement and summed. Scores higher than 36 for women and higher than 38 for men indicate high pain-related fear.
Physical activity and sedentary behavior (self-estimated time, questionnaire) | Participants will complete the questionnaires before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  Self-reported minutes per week or everyday of physical exercise, everyday physical activity and sedentary time.
Body fatness (physiological parameter) | A research assistant will measure each participant before and later at 12-month follow-up of rehabilitation.
  Bioelectrical impedance analysis is used
Body weight (physiological parameter) | A research assistant will measure each participant before and later at 12-month follow-up of rehabilitation
  Using Bioelectrical impedance analysis
Biomarkers explored from blood samples (physiological parameters such as proteins, lipids, metabolites and micro-RNA) | Blood samples will be collected for all participants before, immediately after the rehabilitation (12 weeks) and later at 12-month follow-up.
  The blood samples will be sent to our clinic´s research laboratory to perform exploratory omics analysis, that is, which proteins, metabolites and lipoproteins will be identified cannot be determined in advance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain and Rehabilitation clinic, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Although we received full ethical authorization for this study, we do not have authorization to make the raw data available. Even though data are anonymized, these registry data are still considered sensitive information by the Swedish authorities and restrictions apply to making the data publicly available. The data are available upon request, and data requests should be sent to the Swedish Ethics Committee (registrator@etikprovning.se).

REFERENCES:
- [Background] Gerdle B, Molander P, Stenberg G, Stalnacke BM, Enthoven P. Weak outcome predictors of multimodal rehabilitation at one-year follow-up in patients with chronic pain-a practice based evidence study from two SQRP centres. BMC Musculoskelet Disord. 2016 Nov 25;17(1):490. doi: 10.1186/s12891-016-1346-7. PMID 27887616
- See also: Gerdle B, Rivano Fischer M, Ringqvist A. Interdisciplinary Pain Rehabilitation Programs: Evidence and Clinical Real-World Results. In: Aslanidis T, Nouris C, eds. Pain Management - From Acute to Chronic and Beyond. Rijeka: IntechOpen; 2022: Ch. 2. — http://dx.doi.org/10.5772/intechopen.102411